CLINICAL TRIAL: NCT06918600
Title: The Effect of Exercises for Early Mobilization With Virtual Reality Application on Patients Undergoing Open Heart Surgery
Brief Title: Exercises for Early Mobilization of Patients Undergoing Open Heart Surgery With Virtual Reality Application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yakup Akyüz, research assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: İstanbulU/2025/1
Record Dates: First submitted 2025-02-07; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Early Mobilization, Open-heart Surgery, Virtual Reality
Keywords: virtual reality, open heart surgery, early mobilization, nursing, surgery, postoperative care

STUDY DESIGN:
Intervention Model Description: This study employs a randomized controlled trial (RCT) design to evaluate the effects of virtual reality (VR) applications on early mobilization in patients who have undergone open-heart surgery. The interventional model involves two groups: Intervention Group: Participants in this group will use VR technology to engage in guided mobilization exercises. VR applications will provide structured, engaging, and interactive sessions designed to enhance physical activity and recovery. Each session includes a combination of breathing exercises, lower limb movements, and mobilization strategies presented through a user-friendly VR interface. Control Group: Participants in the control group will receive standard post-operative care, including mobilization as routinely practiced in the clinical setting. No VR application will be used in this group.
Who Masked: Participant
Masking Description: In this study, participants and clinicians administering the intervention will not be masked due to the nature of the virtual reality (VR) application. However, the data analysis will be blinded to ensure unbiased interpretation of results. The analysts will not have access to group allocation information, allowing for objective evaluation of the collected data. No additional parties involved in the clinical trial, beyond the data analysts, are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group: Virtual Reality-Supported Early Mobilization Exercises (Experimental): Participants in this group will use a virtual reality (VR) application designed to support early mobilization after open-heart surgery. The VR application includes guided breathing exercises, lower limb movements, and structured mobilization strategies. These sessions will be conducted using a VR headset, with supervision from a healthcare professional to ensure safety and correct execution.
  Interventions: Other: Virtual Reality-Supported Early Mobilization Program
- Control Group: Standard Postoperative Care and Mobilization (No Intervention): Participants in this group will receive standard postoperative care, including mobilization practices routinely implemented in the clinical setting. This involves assisted physical activity, such as walking and light exercises, guided by the clinical team. No VR intervention will be applied to this group.

INTERVENTIONS:
Other: Virtual Reality-Supported Early Mobilization Program — The intervention involves the use of a virtual reality (VR)-supported mobilization program specifically designed for patients recovering from open-heart surgery. Participants wear a VR headset that delivers guided sessions comprising:
  Breathing Exercises: Deep breathing and coughing techniques to support respiratory function and prevent complications.
  Lower Limb Exercises: Interactive movements aimed at improving circulation and preventing venous stasis.
  Mobilization Strategies: Gradual and guided steps to assist patients in transitioning from bed to ambulation, tailored to their recovery stage.
  This intervention is unique because it integrates an immersive and engaging digital environment to promote physical activity, reduce anxiety, and enhance motivation during the critical early postoperative phase. Unlike standard rehabilitation practices, the VR program provides real-time feedback and visual cues to ensure correct execution of movements.
  Other Names: VR Early Mobilization Program; Virtual Rehabilitation Exercises
  Arms: Intervention Group: Virtual Reality-Supported Early Mobilization Exercises

SUMMARY:
This study aims to evaluate the effectiveness of virtual reality (VR) applications in promoting early mobilization exercises for patients undergoing open-heart surgery. Virtual reality is a non-invasive, easily accessible, and innovative method increasingly used in healthcare settings, including rehabilitation and exercise interventions. Evidence from the literature highlights VR's potential to reduce anxiety, and improve recovery in various patient groups. Despite its extensive applications, there is limited research on the impact of VR in the early postoperative care of cardiac surgery patients. This study addresses this gap by investigating the role of VR-based exercises in improving physical activity and rehabilitation outcomes during the critical early recovery period after surgery. Participants will engage in a VR-supported rehabilitation program during their hospital stay. The study will assess the effects of VR exercises on early mobilization, and overall recovery. The results aim to contribute to the growing field of digital health and provide evidence for integrating VR into postoperative care to enhance the quality of nursing care and patient outcomes.

DETAILED DESCRIPTION:
This study investigates the effectiveness of virtual reality (VR) applications in supporting early mobilization exercises for patients undergoing open-heart surgery. The intervention leverages VR technology as a non-invasive, accessible, and engaging tool to enhance recovery outcomes in the critical early postoperative period. While VR has been widely used in rehabilitation for various patient populations, its application in cardiac surgery for early mobilization remains limited and underexplored. Using a randomized controlled trial design, this research evaluates the impact of VR-based exercises compared to standard care on patients' physical activity, motivation, and recovery. The intervention focuses on promoting physical mobility through interactive VR modules designed to facilitate rehabilitation exercises in a hospital setting. Additionally, the study examines the psychological and social benefits of VR, including its potential to reduce anxiety and improve emotional well-being during the recovery process. This research aims to address a gap in the literature by focusing on the early postoperative phase, where effective mobilization is critical to preventing complications and promoting faster recovery. The study is aligned with the Republic of Turkey's 12th Development Plan, emphasizing the integration of digital health technologies into routine healthcare services to improve patient outcomes and quality of care. The findings from this study are expected to provide valuable evidence supporting the adoption of VR in postoperative care for open-heart surgery patients. By demonstrating its effectiveness as a cost-efficient and scalable intervention, this research seeks to contribute to the development of innovative and patient-centered approaches in nursing care and digital health practices.

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily agreed to participate in the study and written consent was obtained,
* 18 years and over,
* Literate,
* Understand and speak Turkish language,
* No sensory problem (auditory, visual)
* Person, place and time oriented,
* No cognitive problems in expressing themselves,
* Does not have any physical limitation (disability),
* Patients undergoing planned open heart surgery for the first time

Exclusion Criteria:

* Patients with neurological problems (stroke, etc.),
* Patients who develop complications related to surgery in the clinic (delirium, arterial fibrillation, sternal angulation, etc.),
* History of cerebrovascular events,
* Patients with a Glasgow scale <15,
* Patients with complaints of vertigo, dizziness, etc.
* Patients with impaired hemodynamics when wearing glasses
* Deterioration of the general condition of the patient
* Patient abandonment of the study
* Death of the patient
* Patients who develop nausea and vomiting while wearing virtual reality glasses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure: Changes in mobility levels | 1 DAY
  Description: Evaluated using the Patient Mobility Scale to assess patients' ability to perform activities such as sitting, standing, and walking during the early postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: yakup akyüz, research assistant, Principal Investigator — istanbul university faculty of nursing department of surgical diseases nursing
Locations (1):
- Istanbul University, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The following Individual Participant Data (IPD) will be shared as part of this study:
  De-identified Participant Data:
  Demographic and baseline characteristics (age, gender, clinical history). Outcome measures, including mobility scores, pain levels (VAS), kinesiophobia scores (Tampa Scale), walking distance, and step count.
  Length of hospital stay.
  Data Types:
  Primary and secondary outcome data collected during the intervention period.
  Exclusions:
  No personally identifiable information (e.g., names, hospital IDs) will be shared to ensure confidentiality.
  Data Format:
  Data will be shared in anonymized datasets suitable for statistical analysis (e.g., CSV or Excel format).
  This data will be made available to researchers upon request and approval, solely for academic purposes, and in accordance with ethical guidelines and data-sharing agreements.
Supporting Information: SAP, CSR
Time Frame: Start Date: Data will be available starting 6 months after the publication of study results.
  End Date: Data access will remain open for 5 years following the start date. This time frame ensures adequate time for data curation and compliance with ethical and legal guidelines while allowing ample opportunity for secondary research.
Access Criteria: Who Can Access:
  Researchers affiliated with academic, non-profit, or healthcare institutions. Individuals conducting studies for non-commercial purposes.
  What Can Be Accessed:
  De-identified participant-level data, including baseline characteristics and outcome measures.
  Study protocol, statistical analysis plan, and informed consent templates.
  How to Access:
  Researchers must submit a formal data request, including a research proposal, study objectives, and intended use of the data.
  Requests should be directed to the corresponding author or principal investigator via the designated contact email.
  A data-sharing agreement will be required to ensure ethical use, confidentiality, and compliance with applicable regulations.
  Conditions:
  Access will only be granted for projects aligned with the original study objectives or for advancing related scientific knowledge.
  Data must not be shared with third parties or used for commercial purposes. Acknowledgment of the original study in any resu

REFERENCES:
- [Background] Bruno RR, Vlake JH, Molina CA, Aubin H. Editorial: Virtual reality in acute cardiovascular care. Front Cardiovasc Med. 2024 Nov 5;11:1504019. doi: 10.3389/fcvm.2024.1504019. eCollection 2024. No abstract available. PMID 39563940
- [Background] Samant S, Bakhos JJ, Wu W, Zhao S, Kassab GS, Khan B, Panagopoulos A, Makadia J, Oguz UM, Banga A, Fayaz M, Glass W, Chiastra C, Burzotta F, LaDisa JF Jr, Iaizzo P, Murasato Y, Dubini G, Migliavacca F, Mickley T, Bicek A, Fontana J, West NEJ, Mortier P, Boyers PJ, Gold JP, Anderson DR, Tcheng JE, Windle JR, Samady H, Jaffer FA, Desai NR, Lansky A, Mena-Hurtado C, Abbott D, Brilakis ES, Lassen JF, Louvard Y, Stankovic G, Serruys PW, Velazquez E, Elias P, Bhatt DL, Dangas G, Chatzizisis YS. Artificial Intelligence, Computational Simulations, and Extended Reality in Cardiovascular Interventions. JACC Cardiovasc Interv. 2023 Oct 23;16(20):2479-2497. doi: 10.1016/j.jcin.2023.07.022. PMID 37879802
- [Background] Chiu PL, Li H, Yap KY, Lam KC, Yip PR, Wong CL. Virtual Reality-Based Intervention to Reduce Preoperative Anxiety in Adults Undergoing Elective Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2340588. doi: 10.1001/jamanetworkopen.2023.40588. PMID 37906193
- [Background] Rousseaux F, Dardenne N, Massion PB, Ledoux D, Bicego A, Donneau AF, Faymonville ME, Nyssen AS, Vanhaudenhuyse A. Virtual reality and hypnosis for anxiety and pain management in intensive care units: A prospective randomised trial among cardiac surgery patients. Eur J Anaesthesiol. 2022 Jan 1;39(1):58-66. doi: 10.1097/EJA.0000000000001633. PMID 34783683
- [Background] Mendez KJW, Piasecki RJ, Hudson K, Renda S, Mollenkopf N, Nettles BS, Han HR. Virtual and augmented reality: Implications for the future of nursing education. Nurse Educ Today. 2020 Oct;93:104531. doi: 10.1016/j.nedt.2020.104531. Epub 2020 Jul 7. No abstract available. PMID 32711132
- [Background] Chen FQ, Leng YF, Ge JF, Wang DW, Li C, Chen B, Sun ZL. Effectiveness of Virtual Reality in Nursing Education: Meta-Analysis. J Med Internet Res. 2020 Sep 15;22(9):e18290. doi: 10.2196/18290. PMID 32930664